CLINICAL TRIAL: NCT06453798
Title: Effect of Cervical Exercise Combined With Nerve Mobilization on Cervical Spondylotic Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quanzheng Chen (Other)
Responsible Party: Sponsor-Investigator, Quanzheng Chen, Primary rehabilitation therapist, Lingshan County second People's Hospital
Organization: Lingshan County second People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20230601001
Record Dates: First submitted 2024-06-01; First posted 2024-06-12 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Radiculopathy, Cervical
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cervical spine exercises (Experimental): Cervical spine exercise training, patients received the intervention, once a day, 6 times a week, 2 weeks as a course of intervention, a total of 2 courses of intervention
  Interventions: Other: cervical spine exercises
- Neuromobilization (Experimental): Neuromobilization, patients received this intervention, once a day, 6 times a week, 2 weeks as a course of intervention, a total of 2 courses of intervention
  Interventions: Other: Neuromobilization
- cervical spine exercises combined with nerve mobilization (Experimental): cervical spine exercises combined with nerve mobilization，patients received this intervention, once a day, 6 times a week, 2 weeks as a course of intervention, a total of 2 courses of intervention
  Interventions: Other: cervical spine exercises; Other: Neuromobilization

INTERVENTIONS:
Other: cervical spine exercises — Cervical spine exercise training is a method to improve the neck function through the patient's self-exercise.
  Arms: cervical spine exercises; cervical spine exercises combined with nerve mobilization
Other: Neuromobilization — Neuromobilization is a technical technique for rehabilitation therapists to loosen the trapped nerves of patients with professional methods.
  Arms: Neuromobilization; cervical spine exercises combined with nerve mobilization

SUMMARY:
The objective of this clinical trial was to investigate the effects of cervical spine exercises combined with nerve mobilization in patients with radiculopathy.

The main questions it aims to answer are:

1. Whether cervical spine operation combined with nerve mobilization is effective for cervical radiculopathy.
2. Is there any difference between cervical spine operation combined with nerve mobilization and single method? The participants were patients with cervical radiculopathy and were divided into three groups in this study.

1. Experimental group: received cervical spine operation combined with nerve mobilization 2. Control group 1: cervical spine exercises were performed 3. Control group 2: received neuromobilization

DETAILED DESCRIPTION:
After being informed of the risks, participants are required to sign an informed consent form. Eligible participants will be randomly assigned to cervical spine operation combined with nerve mobilizatio or cervical spine exercises or neuromobilization on a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of CSR and have no other complications;
2. Age 18-65 years old, gender unlimited;
3. No other treatment for cervical spondylosis in the last 1 month;
4. No previous surgical treatment for cervical spondylosis;
5. Good compliance;
6. Good mental state, no history of mental illness;
7. Informed consent, and sign the informed consent.

Exclusion Criteria:

1. does not meet the diagnostic criteria;
2. Women during pregnancy;
3. severe stenosis of the foramen;
4. osteoporosis combined with spinal cord tumor, osteomyelitis;
5. infectious diseases, skin defects, allergies;
6. have serious heart, lung and other important organ dysfunction;
7. unable to cooperate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | baseline and 4 weeks
  A scale used to evaluate pain. The scale consists of 0 to 10 points, with a higher score indicating greater pain and a lower one.
Range of motion | baseline and 4 weeks
  The range of motion of the associated joints in the neck was measured using a joint protractor
Muscle strength | baseline and 4 weeks
  The microFET2 instrument was used to test the muscle strength of the neck related muscles.

SECONDARY OUTCOMES:
Tanaka Yasuhisa Cervical Spondylopathy Symptom Scale | baseline and 4 weeks
  To assess the status of the patient's cervical spine. The scale includes a score of -2 to 20, with the larger the score, the less severe the symptoms associated with the cervical spine.
neck disability index. The total score ranges from 0 (accessibility) to 50 (total paralysis), with higher scores indicating more severe dysfunction. | baseline and 4 weeks
  A scale used to assess the degree of cervical spine dysfunction
the medical outcomes study 36-item short-form health survey | baseline and 4 weeks
  A scale used to assess quality of life.The exact score of the SF-36 varies from item to item, but in general, the higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lingshan County second People's Hospital, Qinzhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: No